CLINICAL TRIAL: NCT00323011
Title: A Randomized Pilot Study of the Activation of the Hemostatic Pathway by FOLFIRI + Bevacizumab With or Without Dalteparin in First Line Treatment of Advanced Colorectal Cancer
Brief Title: FOLFIRI + Bevacizumab With or Without Dalteparin in First Line Treatment of Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: drug not available
Sponsor: University of Southern California (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Syma Iqbal, MD, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 3C-05-2
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Dalteparin; Fluorouracil; Leucovorin; Irinotecan; Bevacizumab

ARMS (3):
- Arm A: 5-FU/LV/CPT-11/Bevacizumab (Active Comparator): 5-FU 400 mg/m2, days 1, 15, & 29 Leucovorin Calcium 200 mg/m2, days 1, 15, & 29 CPT-11 180 mg/m2, days 1, 15 & 29 Bevacizumab 5mg/kg, days 1, 15, & 29
  Interventions: Drug: Fragmin, 5-Fluorouracil, Folinic Acid, irinotecan, bevacizumab
- Arm B: 5-FU/LV/CPT-11/Bevacizumab + Dalteparin (Experimental): 5-FU 400 mg/m2, days 1, 15, & 29 5-FU 2400 continuous infusion days 1-2, 15-16, 29-30. Leucovorin Calcium 200 mg/m2, days 1, 15, & 29 CPT-11 180 mg/m2, days 1, 15 & 29 Bevacizumab 5mg/kg, days 1, 15, & 29 Dalteparin 5000 IU subcutaneous starting cycle 2, days 1, 15, & 29
  Interventions: Drug: Fragmin, 5-Fluorouracil, Folinic Acid, irinotecan, bevacizumab
- 5-FU/LV/CPT-11/Bevacizumab+Dalteparin daily (Experimental): 5-FU 400 mg/m2, days 1, 15, & 29 5-FU 2400 continuous infusion days 1-2, 15-16, 29-30. Leucovorin Calcium 200 mg/m2, days 1, 15, & 29 CPT-11 180 mg/m2, days 1, 15 & 29 Bevacizumab 5mg/kg, days 1, 15, & 29 Dalteparin 5000 IU subcutaneous starting cycle 2, daily
  Interventions: Drug: Fragmin, 5-Fluorouracil, Folinic Acid, irinotecan, bevacizumab

INTERVENTIONS:
Drug: Fragmin, 5-Fluorouracil, Folinic Acid, irinotecan, bevacizumab

SUMMARY:
This study is for people with colorectal cancer, who have tumors that cannot be completely removed by surgery. Blood clots are a problem in patients with cancer. Blood clots are also a problem in patients receiving cancer drugs. Studies have shown that up to 17% of patients receiving cancer drugs experienced blood-clotting problems. One purpose of this study is to find if the drug combination of irinotecan, 5-fluorouracil (5-FU), bevacizumab and leucovorin (LV) affect blood-clotting factors. A second purpose of this study is to find out what effects the drug dalteparin has on clotting factors in the blood in patients receiving the drug combination of irinotecan, 5-FU, bevacizumab and LV. It is hoped that adding dalteparin to chemotherapy may benefit patients with colorectal cancer by preventing blood clots

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed metastatic or recurrent colorectal tumors with no previous treatment for advanced disease.
* Age > 18 years (as no dosing or toxicity data are currently available on the use of 5-FU/CPT11 + bevacizumab + dalteparin in patients <18 years of age).
* SWOG performance status 0-1.
* Patients must have adequate organ and marrow function as defined below, with tests performed no more than seven days prior to the first study drug administration:leukocytes >3.0, absolute neutrophil count >1,500/ml,platelets > 100 X 109 L ,total bilirubin < upper normal institutional limits,AST(SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal ( or < 5x the upper normal institutional limits in the case of liver metastases,alkaline phosphatase < 2.5 X institutional upper limit of normal ( or < 5x the upper normal institutional limits in the case of liver metastases or < 10x the upper normal institutional limits in the case of bone disease, Serum creatinine < 1.6 mg/dL OR Calculated creatinine clearance > 40 mL/min/1.73 m2, PT, PTT, within normal range, Urine protein/creatinine ratio < 1.0
* At least one measurable lesion according to the RECIST criteria which has not been irradiated (i.e. newly arising lesions in previously irradiated areas are accepted). Ascites, pleural effusion, and bone metastases are not considered measurable. Minimum indicator lesion size: > 10 mm measured by spiral CT or >20mm measured by conventional techniques.
* The effects of chemotherapy on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study participation and 30 days from the date of the last study drug administration (postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential). Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and willingness to sign a written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
* Have a negative serum pregnancy test within 7 days prior to initiation of chemotherapy (female patients of childbearing potential).
* Life expectancy of at least 12 weeks.
* Fully recovered from any surgical procedure

Exclusion Criteria:

* Lactating woman unwilling to stop breast feeding for the duration of study participation and 30 days from the date of the last study drug administration
* History of allergy to any of the chemotherapeutics or antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy.
* Prior unanticipated severe reaction to fluoropyrimidine therapy, known hypersensitivity to 5-fluorouracil, or known DPD deficiency.
* Serious, uncontrolled, intercurrent infection(s) or illnesses including, but not limited to ongoing or active infection, symptomatic congestive heart failure, or unstable angina pectoris, or cardiac arrhythmia.
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer.
* Current, recent (within 4 weeks of first infusion on this study) or planned participation in an investigational drug study.
* Patients with documented DIC (disseminated intravascular coagulation).
* Patients with a previous history of a bleeding diathesis or significant bleeding episode such as gastrointestinal bleeding or a CNS hemorrhage.
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) within the last 12 months.
* Presence of central nervous system or brain mets.
* Major surgery, open biopsy, or significant traumatic injury within 28 days prior to Day 1, or anticipation of need for major surgical procedure during the course of the study.
* Unwillingness to participate or inability to comply with the protocol for the duration of the study.
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 1.
* Blood pressure > 150/100 mmHg.
* Unstable angina.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of myocardial infarction or stroke within 6 months.
* Clinically significant peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* History of abdominal fistula, gastrointestinal perforation or intrabdominal abscess within 28 days prior to Day 0.
* Serious, non-healing wound, ulcer or bone fracture.
* Carcinoma of any histology in close proximity to a major vessel, lung cavitation or history of hemoptysis.
* Completion of previous chemotherapy regimen < four weeks prior to the start of study treatment (within six weeks of study treatment for mitomycin C and nitrosureas), or with related toxicities unresolved prior to the start of study treatment.
* Patients who are taking anti coagulation therapy such as coumadin or low molecular weight Heparin.
* Patients who have an allergy against heparin.
* Medical, social or psychological factors which would interfere with consent and follow up.
* Known defective hemostasis, e.g. thrombocytopenia.
* Patients receiving Hormone Replacement Therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-05; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, MD, Principal Investigator — University of Southern California
Locations (1):
- USCNorris Hospital, Los Angeles, California, United States